CLINICAL TRIAL: NCT05635058
Title: Effect of Reminiscence Therapy on Functioning of Older Adults: A Randomized Controlled Study
Brief Title: Effect of Reminiscence Therapy on Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Done Gunay, PhD student, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TELGUNAY1
Record Dates: First submitted 2022-11-10; First posted 2022-12-02 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Nurse's Role
Keywords: reminiscence therapy; functionality; nursing; older adults; care

STUDY DESIGN:
Intervention Model Description: The study was conducted as the randomized controlled experimental trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminisence Therapy (Experimental): The participants in the intervention group received reminiscence therapy which was implemented by the researcher as one session per week for eight weeks. In the reminiscence sessions, mnemonic materials selected specifically for the determined interview topic were used. In the sessions, topics such as childhood life, work life, religious holidays, national holidays, old songs, military ceremonies, wedding ceremonies, gardening and field work were shared. In the reminiscence sessions, the participants were encouraged to verbally express the feelings and thoughts they remembered about the mnemonics. The interviews were recorded by the researcher and each session lasted 45-60 minutes. At the end of the reminiscence session, the topics addressed in the session were summarized by the researcher.
  Interventions: Other: The Reminisence Therapy
- Control Group (No Intervention): Interviews were conducted with the individuals in the control group on a designated day of the week, at a designated place in the nursing home. The researcher interviewed the individuals in the control group once a week for eight weeks. During these meetings, daily issues and events such as health, sports, and weather were discussed. Each of the mentioned interviews lasted 45-60 minutes. At the end of eight weeks, SMMT and the "Multidimensional Observation Scale for Elderly Individuals" were implemented again to the participants in the intervention and control groups.

INTERVENTIONS:
Other: The Reminisence Therapy — Reminiscence sessions were held in a meeting room in the nursing home and arranged in accordance with the interviews. In the reminiscence sessions, mnemonic materials selected specifically for the determined interview topic were used. The materials to be used in the reminiscence sessions were determined in accordance with the education level and cultural characteristics of the participants. In the sessions, topics such as childhood life, work life, religious holidays, national holidays, old songs, military ceremonies, wedding ceremonies, gardening and field work were shared. In the reminiscence sessions, the participants were encouraged to verbally express the feelings and thoughts they remembered about the mnemonics. The interviews were recorded by the researcher and each session lasted 45-60 minutes. At the end of the reminiscence session, the topics addressed in the session were summarized by the researcher, the following weeks topic was determined and the interview was concluded.
  Arms: Reminisence Therapy

SUMMARY:
This study was conducted to examine the effect of reminiscence therapy on the functionality of older adults aged 65 and over living in nursing homes.

DETAILED DESCRIPTION:
ABSTRACT Objective : This study was conducted to examine the effect of reminiscence therapy on the level of functionality of individuals aged 65 and over.

Method: The sample of the study consisted of 16 residents who lived in a public nursing home between December 2019 and February 2020 and agreed to participate in the study. Participants were divided into intervention and control groups using the simple random sampling method. Reminiscence therapy was performed with each participant in the intervention group for 8 weeks. The participants in the control group received routine services and were regularly visited for 8 weeks. The research data were obtained by implementing the "Personal Information Form," "Multidimensional Observation Scale for Elderly Subjects (MOSES), and "Mini Mental State Examination (MMSE)" with all participants before the reminiscence therapy and at the end of week eight. Non-parametric tests were completed in analyzing the data as the sample size was lower than 30.

Findings: It was determined that 87.5% of the participants in the intervention group had a chronic disease, 50% were male, and 37.5% were elementary school graduates. All the participants in the control group had a chronic disease, 62.5% were male, and 50% were elementary school graduates. When the pre- and post-reminiscence therapy results were compared, a significant difference was found in the MMSE and MOSES (in the areas of disoriented behavior, depressed/anxious mood, and withdrawn behavior) scores in the intervention group. In the post-test evaluation, a significant difference was found between the intervention and comparison group in MOSES scores. It was determined that the participants in the intervention group that received reminiscence therapy had better functional and cognitive competency than the control group in the areas of self-care, depression/anxiety, and withdrawal from society.

Conclusion: It was concluded that the reminiscence therapy contributed to increase the mental competence and functionality of the older adult participants.

ELIGIBILITY:
Inclusion Criteria:

* were 65 years of age and older
* had a Standardized Mini Mental Test (SMMT) score between 24 and 30
* Individuals who did not have communication difficulties and mental problems
* agreed to participate in the study were included in the study sample.

Exclusion Criteria:

* were 64 years of age and younger
* have communication difficulties and mental problems
* had a Standardized Mini Mental Test (SMMT) score 24 and more less
* nor agreed to participate in the study.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Standardized Mini-Mental State Exam (MMSE): | 5 minutes
  Developed by Folstein et al., SMMT is a short, useful, and standardized assessment tool that can be used to determine the cognitive level globally. The test consists of five subsections: orientation of time and space, recording memory, attention, recall, and language. MMSE can be applied by physicians, nurses, and psychologists in a short time. The highest score that can be obtained in MMSE is 30. In the test, a score of 24-30 points is considered normal, 20-23 mild dementia, 10-19 moderate dementia, and 0-9 advanced dementia (Folstein et al. 1975). The validity and reliability study of the test for Turkish population was completed by Güngen et al. (2002).
Multidimensional Observation Scale for Elderly Subjects (MOSES): | 15 minutes
  MOSES is a multi-dimensional measurement tool developed by Helmes, Csapo, and Short to evaluate the functionality of older adults (Helmeset al., 1987). The scale consists of 40 questions and provides evaluation in 5 functional sub-dimension areas. The dimensions of the scale are Self-Care , Disorientation , Depressed/Anxious Mood, Irritable behavior, and Withdrawal from society. Each item in the scale is scored between 0 and 4. Twenty-two items of the scale have 4 choices and 18 items have 5 choices. The last option in the five-choice items was created with the thought that the older adult would not be able to answer the question and/or the question would not be suitable for the older adult. The lowest score that can be obtained from the scale is 0, and the highest score is 138. A low score indicates that the functionality of the older adult is high, while a high score indicates that the functionality of the older adult is low (Helmes et al. 1987).

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet Univercity, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Shropshire M. Reminiscence intervention for community-dwelling older adults without dementia: a literature review. Br J Community Nurs. 2020 Jan 2;25(1):40-44. doi: 10.12968/bjcn.2020.25.1.40. PMID 31874077
- [Background] Westerhof GJ, Bohlmeijer ET. Celebrating fifty years of research and applications in reminiscence and life review: state of the art and new directions. J Aging Stud. 2014 Apr;29:107-14. doi: 10.1016/j.jaging.2014.02.003. Epub 2014 Mar 13. PMID 24655678
- [Background] Henkel LA, Kris A, Birney S, Krauss K. The functions and value of reminiscence for older adults in long-term residential care facilities. Memory. 2017 Mar;25(3):425-435. doi: 10.1080/09658211.2016.1182554. Epub 2016 May 10. PMID 27161334
- [Background] Kris AE, Henkel LA. Remembering Reminiscence. J Gerontol Nurs. 2017 Jun 1;43(6):3-4. doi: 10.3928/00989134-20170512-01. No abstract available. PMID 29975785
- [Background] Wong PT, Watt LM. What types of reminiscence are associated with successful aging? Psychol Aging. 1991 Jun;6(2):272-9. doi: 10.1037//0882-7974.6.2.272. PMID 1863396
- [Background] Stinson CK. Structured group reminiscence: an intervention for older adults. J Contin Educ Nurs. 2009 Nov;40(11):521-8. doi: 10.3928/00220124-20091023-10. PMID 19904866
- [Background] King DB, Cappeliez P, Canham SL, O'Rourke N. Functions of reminiscence in later life: Predicting change in the physical and mental health of older adults over time. Aging Ment Health. 2019 Feb;23(2):246-254. doi: 10.1080/13607863.2017.1396581. Epub 2017 Nov 7. PMID 29110517